CLINICAL TRIAL: NCT01077830
Title: A Multinational, Observational Follow-Up Study of the Incidence of Cancer and Mortality in Patients From the SEAS Trial
Brief Title: An Observational Follow-Up Study of the Incidence of Cancer and Mortality in Patients From the SEAS (Simvastatin and Ezetimibe in Aortic Stenosis) Trial (MK-0653A-043-10)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Collaborators: Institute of Applied Economics Aps, Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0653A-043-10; 2010_016 (Other: Merck Registration Number)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: New Incidence of Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ezetimibe/Simvastatin 10/40 mg: Participants who received Ezetimibe/Simvastatin 10/40 mg in the base study
- Placebo: Participants who received placebo in the base study

SUMMARY:
The purpose of this extension is to observe the incidence rates of cancer, total mortality, and mortality due to cancer over a 21 month follow-up period in patients from the SEAS trial (2004_050, MK0653A-043; NCT00092677).

DETAILED DESCRIPTION:
The SEAS Follow-up Study is a 21 month extension to the base protocol (2004_050, MK0653A-043; NCT00092677). The main objective of the extension is to observe the incidence rates of cancer, total mortality, and mortality due to cancer over a 21 month follow-up period (from 04-March 2008 to 31-December 2009) in patients from the SEAS clinical trial. The sources of study data will include data collected from national cancer and death registries as well as data from the original clinical trial. No patient visits will occur. National cancer and death registries exist in 5 of the 7 countries that participated in the base SEAS trial. At the time of Follow-up study initiation, accessing the registry data in Ireland was not feasible due to local regulations and Cancer and Death registries did not exist in Germany. As a result, data will be collected only for all SEAS patients known to be alive at the end of the base study originating from Sweden, Denmark, Norway, Finland, and the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* The cohort will include all patients from the five participating countries (Sweden, Denmark, Norway, Finland, and United Kingdom) who were randomized into the SEAS base study and who were known to be alive at the end of the base study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will include all patients from the five participating countries (Sweden, Denmark, Norway, Finland, and United Kingdom) who were randomized into the SEAS base study and who were known to be alive at the end of the base study.
Sampling Method: Non-Probability Sample
Enrollment: 1392 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Green A, Ramey DR, Emneus M, Iachina M, Stavem K, Bolin K, McNally R, Busch-Sorensen M, Willenheimer R, Egstrup K, Kesaniemi YA, Ray S, Basta N, Kent C, Pedersen TR. Incidence of cancer and mortality in patients from the Simvastatin and Ezetimibe in Aortic Stenosis (SEAS) trial. Am J Cardiol. 2014 Nov 15;114(10):1518-22. doi: 10.1016/j.amjcard.2014.08.016. Epub 2014 Aug 27. PMID 25267716
- See also: Current view of trial on ClinicalTrials.gov — http://www.clinicaltrials.gov/ct2/show/NCT00092677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants from five countries (Sweden, Denmark, Norway, Finland, and United Kingdom) who completed the SEAS base study and who were known to be alive at the end of the base study.
Pre-assignment Details: Of the 1873 participants in the SEAS base study, 1392 were eligible for inclusion in this follow-up study. Of these 1392 participants, 33 were excluded due to incomplete base study data or because follow-up data could not be obtained, leaving 1359 participants in the follow-up study.
Groups:
- Placebo: Participantss who received placebo in the base study
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo
Started | 677 | 682
Completed | 677 | 682
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo | Total
Number analyzed (Participants) | 677 | 682 | 1359
Age, Customized [Number; unit: Participants]
  < 50 years | 4 | 3 | 7
  50 to 59 years | 92 | 91 | 183
  60 to 69 years | 160 | 189 | 349
  70 to 79 years | 250 | 234 | 484
  ≥80 years | 171 | 165 | 336
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 272 | 539
  Male | 410 | 410 | 820

OUTCOME MEASURES:

1. Secondary Outcome: Crude Rate of Death (Any Cause) - Follow-up Total Cohort
Description: All deaths reported during follow-up were reviewed by the Expert Review Committee to ascertain cause of death. The crude rates of death for each arm were calculated as follows: Number of participants in the arm was multiplied by the Duration of Follow-up (days) and divided by 365 (days per year) to establish the Total Participant-years for the arm. The Number of Deaths (any cause) reported was divided by the Total Participant-years and the resultant quotient was then multiplied by 100 to determine the Rate of Death.
Time Frame: up to 21 Months after the end of the base study
Population: Primary analysis population was Follow-Up Total Cohort defined as all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: per 100 participant-years
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo
Number analyzed (Participants) | 677 | 682
per 100 participant-years | 3.59 [2.67 to 4.85] | 2.70 [1.92 to 3.80]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 mg vs Placebo; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.84 to 2.09] — Hazard Ratio obtained by dividing the crude rate of death (any cause) reported in the Ezetimibe/Simvastatin 10/40 arm by the crude rate of death (any cause) in the Placebo arm

2. Secondary Outcome: Crude Rate of Death Due to Cancer - Follow-up Primary Cohort
Description: All deaths reported during follow-up were reviewed by the Expert Review Committee to ascertain if cancer was cause of death. The crude rates of death due to cancer for each arm were calculated as follows: Number of participants in the arm was multiplied by the Duration of Follow-up (days) and divided by 365 (days per year) to establish the Total Participant-years for the arm. The Number of Deaths due to Cancer reported was divided by the Total Participant-years and the resultant quotient was then multiplied by 100 to determine the Crude Rate of Death Due to Cancer.
Time Frame: up to 21 Months after the end of the base study
Population: Analysis population was Follow-up Primary Cohort defined as all participants in the follow-up study without a history of cancer before the start of the follow-up period.
Measure: Number (95% Confidence Interval); unit: per 100 participant-years
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo
Number analyzed (Participants) | 595 | 599
per 100 participant-years | 0.38 [0.14 to 1.01] | 0.28 [0.09 to 0.86]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.30 to 6.06] — Hazard Ratio obtained by dividing the crude rate of death from cancer reported in the Ezetimibe/Simvastatin 10/40 arm by the crude rate of death from cancer in the Placebo arm

3. Primary Outcome: Crude Rate of Newly Diagnosed Cancer-Follow-up Primary Cohort
Description: Any incidence of cancer reported during follow-up that was assessed by the Expert Review Committee to be a new case of cancer. The crude new cancer rates for each arm were calculated as follows: Number of participants in the arm was multiplied by the Duration of Follow-up (days) and divided by 365 (days per year) to establish the Total Participant-years for the arm. The Number of New Cancers reported was then divided by the Total Participant-years and the resultant quotient was then multiplied by 100 to determine the Crude New Cancer Rate.
Time Frame: up to 21 Months after the end of the SEAS (base) study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: per 100 participant-years
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo
Number analyzed (Participants) | 595 | 599
per 100 participant-years | 1.14 [0.65 to 2.01] | 2.07 [1.36 to 3.15]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/40 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.27 to 1.11] — Hazard Ratio obtained by dividing the crude rate of new cancers reported in the Ezetimibe/Simvastatin 10/40 arm by the crude rate of newly diagnosed cancers in the the Placebo arm

ADVERSE EVENTS:
Description: No formal reporting or recording of adverse events was conducted during this observational study
Groups:
- Ezetimibe/Simvastatin 10/40 mg: Participants who were assigned to the Ezetimibe/Simvastatin 10/40 mg cohort in the base study
- Placebo: Participants who were assigned to the placebo cohort in the base study
Arm/Group | Ezetimibe/Simvastatin 10/40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.